CLINICAL TRIAL: NCT00170573
Title: Comparison of Quality of Life in Patients With Platinum-sensitive Recurrent Ovarian, Fallopian Tube and Peritoneal Cancer When Treated With Treatment With Trabectedin/PLD or Standard Platinum-based Therapy
Brief Title: Caelyx Biweekly in Heavily Pretreated Patients With Relapsed Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: North Eastern German Society of Gynaecological Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Noggo ov4
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Results first posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-11

CONDITIONS: Ovarian Cancer
Keywords: Pegylated liposomal doxorubicin; PPE; Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Caelyx (Experimental): 40 mg/m² biweekly
  Interventions: Drug: Caelyx

INTERVENTIONS:
Drug: Caelyx — 40 mg/m² biweekly

SUMMARY:
Effect of biweekly schedule of PLD on dose-limiting toxicity of PPE and patient's quality of life

DETAILED DESCRIPTION:
Pegylated liposomal doxorubicin (PLD) formulation has been approved for the treatment of recurrent ovarian cancer (ROC). Toxic skin reactions e.g. palmar-plantar erythrodysesthesia (PPE) were reported as being the dose-limiting toxicity and have an impact on patients' quality of life (QoL). The primary aim of this study was to optimise the toxicity profile by choosing a biweekly schedule of PLD Furthermore, QoL was investigated. Secondary objective of this study was to evaluate the response rates of this new regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age
* recurrent ovarian, peritoneal, or tubal cancer and prior treatment with platinum- and paclitaxel were eligible to this trial.
* Eastern Cooperative Oncology Group (ECOG) performance status less than 3.
* renal function (serum creatinine 1.25 times the upper limit of normal, glomerular filtration rate greater than 60 ml/min)
* liver function (AST/ ALT three times the upper limit of normal, bilirubin concentrations 1.25 the upper limit of normal)
* bone marrow function (neutrophil count greater than 1.5 x 109/l, and a platelet count greater than 100 x 109/l).

Exclusion Criteria:

* patients with more than 4 chemotherapies in medical history
* severe cardiac disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2001-09; Primary Completion 2009-04 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jalid Sehouli, Principal Investigator — Charite University, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment period: September 2001 - February 2004
Period: Overall Study
Arm/Group | Caelyx
Started | 77
Completed | 64
Not Completed | 13
Not completed — Violation of inclusion criteria | 13

BASELINE CHARACTERISTICS:
Groups:
- Caelyx: Caelyx: Caelyx 40 mg/ m2biweekly
Arm/Group | Caelyx
Number analyzed (Participants) | 64
Age, Continuous [Median (Full Range); unit: years] | 59 [38 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 0
Region of Enrollment [Number; unit: participants]
  Germany | 64
Classification of tumour (according to FIGO ovarian cancer staging) [Number; unit: participants] — IA - Tumor limited to one ovary, IB - Tumor limited to both ovaries, IC - Tumor involves 1 or both ovaries + capsule rupture, tumor on surface or positive washings/ascites, IIA - Extension and/or implants on the uterus and/or tube(s), IIB - Extension to other pelvic intraperitoneal tissues, IIC - IIA or IIB with positive washings/ascites, IIIA - Microscopic peritoneal metastasis beyond the pelvis, IIIB - Macroscopic, extrapelvic, peritoneal metastasis ≤ 2 cm, IIIC - Macroscopic, extrapelvic, peritoneal metastasis > 2 cm and/or regional lymph node metastasis, IV - Distant metastasis
  participants
    stage IA | 2
    stage IB | 0
    stage IC | 1
    stage IIA | 8
    stage IIB | 2
    stage IIC | 4
    stage IIIA | 2
    stage IIIB | 3
    stage IIIC | 34
    stage IV | 7
    unknown | 1
Histological grade [Number; unit: participants] — grade 1 - well differentiated; grade 2 - moderately differentiated; grade 3 - poorly differentiated; grade 4 - undifferentiated
  Lower grade tumours generally grow more slowly and are less likely to spread and metastasize than higher grade tumours.
  participants
    grade 1 | 8
    grade 2 | 20
    grade 3 | 28
    grade 4 | 0
    unknown | 8
ECOG performance status [Number; unit: participants] — 0 - Fully active, able to carry on all pre-disease performance without restriction; 1 - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2 - Ambulatory and capable of all selfcare but unable to carry out any work activities, up and about more than 50% of waking hours; 3 - Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours; 4 - Completely disabled; cannot carry on any selfcare; totally confined to bed or chair; 5 - Dead
  participants
    0 | 20
    1 | 34
    2 | 10
    3 | 0
    4 | 0
    5 | 0

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Palmar-plantar Erythrodysesthesia (PPE)
Description: The outcome will be measured by number of participants with reported skin toxicity PPE of CTC (Common Toxicity Criteria)-Grade I / II / III / IV.
  Grade I - Dysesthesia/paraesthesia tingling of hands and feet; Grade II - Discomfort in holding objects and upon walking, painless swelling and erythema; Grade III - painful erythema and swelling of palms and soles, periungual erythema and swelling; Grade IV - Desquamation, ulceration, blistering, severe pain
Time Frame: through study completion, an average of 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Caelyx
Number analyzed (Participants) | 64
Participants
  CTC-Grade I | 18
  CTC-Grade II | 9
  CTC-Grade III | 3
  CTC-Grade IV | 0
  no PPE | 34

2. Secondary Outcome: Overall Survival
Description: Overall survival estimated by the Kaplan-Meier method
Time Frame: for up to 3 years
Measure: Median (Full Range); unit: months
Arm/Group | Caelyx
Number analyzed (Participants) | 64
months | 18.2 [1.4 to 34.0]

ADVERSE EVENTS:
Time Frame: through study completion, an average of 18 months
Description: Patients were asked at each visit for the occurrence of adverse events. Furthermore blood samples for hematological and clinical chemistry assessment were taken at defined time points.
Arm/Group | Caelyx
Serious Adverse Events (participants affected / at risk) | 4/64
Other Adverse Events (participants affected / at risk) | 60/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Caelyx (N=64)
Anemia (Blood and lymphatic system disorders) | 3
Thrombopenia (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Caelyx (N=64)
Leucopenia (Blood and lymphatic system disorders) | 26
PPE (Skin and subcutaneous tissue disorders) | 30
Thrombopenia (Blood and lymphatic system disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No